CLINICAL TRIAL: NCT05260476
Title: To Investigate the Effect of Rreablement Service of Long-term Care on Physical Mobility and Quality of Life in Disable People
Brief Title: The Effect of Reablement Service of Long-term Care on Physical Mobility and Quality of Life in Disable People
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Jia-Ching Chen, c123010@yahoo.com.tw, Tzu Chi University
Other Study IDs: IRB110-277-B
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Reablement; Home Rehabilitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reablement group: The home reablement program will be implemented by a physical therapist according to "Long-term Care Reablement Operational Guidelines" announced by the Ministry of Health and Welfare of Taiwanese government
  Interventions: Other: Reablement
- Non-reablement group: This group will only receive general home care service without the reablement program.
  Interventions: Other: Reablement

INTERVENTIONS:
Other: Reablement — The service provider customizes a training plan and formulates training goals based on the patient's level of disability, family environment, and the needs of the patient and the caregiver.

SUMMARY:
The long-term care 2.0 policy has been launched at 2017 by Taiwanese government to respond the rate of aging population reached to14% and estimated to 20% in 2025, becoming a "super-aged society" in Taiwan. As aging society, the ratio of chronic disease and disability has reasonably raised. The home reablement and care of this policy are not only to prevent and delay disability but provide daily care for the elderly who needed. As the implementation of the policy, there is still insufficient research to investigate and compare the effects on physical mobility and quality of life among the individual after using these different types of the service. Therefore, the aim of the study is to compare the effects on physical function and quality of life of the frail and disabled individual with and without receiving the home reablement services.

The participants will be enrolled from the long-term care service units registered in local government at Hualien county, Taiwan. The recruited participants will be assigned to two groups in a convenient method (receiving and non-receiving the home reablement service). All participants will be assessed by a professional physical therapist at three time points, before the reablement, at 1-3 months after receiving the reablement, then follow-up after 3 months

ELIGIBILITY:
Inclusion Criteria:

* Aged from 50-90 years old
* Be able to follow the command and cooperate with the assessor
* The disability grade level 2 to 8 according to the grading with long-term care case-mix system, approximately to 20 to 80 of Barthel Index score.
* Receiving the reablement services at least 3 times/a set.

Exclusion Criteria:

* Using the outpatient rehabilitation service during the study period
* Transferring or delivering to institution
* Re-admission to hospital during using the service

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Aged from 50-90 years old
  * The disability grade level 2 to 8 according to the grading with long-term care case-mix system, approximately to 20 to 80 of Barthel Index score.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery, SPPB | 15 minutes
  The SPPB is one of the most commonly used instruments for measuring physical performance in population studies of aging. The SPPB consists of three subtests: a hierarchical test of balance, a short walk at usual pace and standing up from a chair five times consecutively. Low scores on the SPPB have a high predictive value for a wide range of health consequences including disability in Activities of Daily Living.

SECONDARY OUTCOMES:
Barthel index, BI | 10 minutes
  The total score is from 0 to 100, each item is divided into 2-4 levels according to complete independence, need assistance and complete dependence. The lower the score, the higher the dependent level.
Instrumental Activities of Daily Living, IADL | 5 minutes
  There are eight domains of function measured with the Lawton IADL scale. Evaluators are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
EuroQol Five Dimensions Questionnaire, EQ-5D | 5 minutes
  The quality of life was assessed using 5 items: Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression. This questionnaire asks respondents to choose the option that best suits them based on their health status.
Elderly Mobility Scale, EMS | 15 minutes
  The EMS is a 7-item objective measure designed to assess mobility and function in elderly adults. Divided into bedside mobility and functional mobility (lying to sitting, sitting to lying, standing, and balance and walking). The total score is 0 to 20 points. The higher the score, the better performance.
Handheld dynamometer to measure muscle strength | 5 minutes
  Grip strength will be measured twice on the left and right sides of the elderly in a standard sitting position with elbow 90 degree and shoulder in neutral position, and the average value will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Ching Chen, Principal Investigator — Department of physical therapy, Tzu Chi University; Lian-Cing Yan, Study Director — Department of physical therapy, Tzu Chi University

IPD SHARING:
Plan to Share IPD: No